CLINICAL TRIAL: NCT04680988
Title: A Randomized,Open-label, Multi-Center, Phase II Clinical Trial to Assess the Efficacy and Safety of SHR-1210± SHR-1020 Versus Physician's Choice Chemotherapy in the Treatment of Recurrent or Metastatic Cervical Cancer Patients
Brief Title: A Study of SHR-1210± SHR-1020 Versus Chemotherapy in Patients With Recurrent or Metastatic Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-II-217
Record Dates: First submitted 2020-12-07; First posted 2020-12-23 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Recurrent or Metastatic Cervical Cancer
MeSH Terms: conditions — Recurrence; Uterine Cervical Neoplasms | interventions — camrelizumab; famitinib; Albumin-Bound Paclitaxel; Pemetrexed; Injections; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Doublet Arm (Experimental): SHR-1210+SHR-1020
  Interventions: Drug: SHR-1210; Drug: SHR-1020
- Single Arm (Experimental): SHR-1210
  Interventions: Drug: SHR-1210
- Physician's choice chemotherapy (Active Comparator): Albumin-bound paclitaxel injection or Pemetrexed disodium for injection or Gemcitabine for injection
  Interventions: Drug: Physician's choice chemotherapy

INTERVENTIONS:
Drug: SHR-1210 — SHR-1210 intravenously every 3 weeks
  Other Names: Camrelizumab
  Arms: Doublet Arm; Single Arm
Drug: SHR-1020 — SHR-1020 Orally once daily
  Other Names: Famitinib
  Arms: Doublet Arm
Drug: Physician's choice chemotherapy — Investigators will declare one of the following regimens:Albumin-bound paclitaxel injection, Pemetrexed disodium for injection, Gemcitabine for injection
  Other Names: Albumin-bound paclitaxel injection, Pemetrexed disodium for injection, Gemcitabine for injection
  Arms: Physician's choice chemotherapy

SUMMARY:
This is a randomized, open-label, 3-arm Phase 2 study to evaluate the efficacy and safety of SHR-1210 alone or with SHR-1020 versus physician's choice chemotherapy in recurrent or metastatic cervical cancer patients. All enrolled patients will be randomly divided into 3 groups and receive treatment until disease progression, intolerable toxicity，any criterion for stopping the study drug or SHR-1210 treatment for up to 2 years.

DETAILED DESCRIPTION:
This is a randomized, open-label, 3-arm Phase 2 study to evaluate the efficacy and safety of SHR-1210 alone or with SHR-1020 versus physician's choice chemotherapy in recurrent or metastatic cervical cancer patients. All enrolled patients will be randomly divided into 3 groups and receive treatment until disease progression, intolerable toxicity，any criterion for stopping the study drug or SHR-1210 treatment for up to 2 years.The primary study hypotheses are that the combination of SHR-1210 plus SHR-1020 is superior to SHR-1210 or physician's choice chemotherapy with respect to: 1) Progression free survival(PFS) in recurrent or metastatic cervical cancer patients(SHR-1210+SHR-1020 versus SHR-1210；2) Overall survival(OS) in recurrent or metastatic cervical cancer patients(SHR-1210+SHR-1020 versus Physician's choice chemotherapy).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily agree to participate by giving written informed consent.
2. Histologically or cytologically confirmed diagnosis of squamous-cell carcinoma, adenosquamous carcinoma, or adenocarcinoma of the cervix.
3. The patients relapsed after a platinum-based treatment regimen for recurrent or metastatic disease.
4. Patients must provide a fresh biopsy. If not, sufficient and adequate tumor tissue sample from the most recent biopsy of a tumor lesion will be required for PD-L1 expression.
5. Has measurable lesion on imaging based on RECIST version 1.1.
6. Have a life expectancy of at least 3 months.
7. ECOG performance status 0-1.
8. If childbearing potential, female patients must be willing to use at least 1 adequate barrier methods throughout the study, starting with the screening visit through 6 months after the last dose of study treatment.

Exclusion Criteria:

1. Has any malignancy <5 years prior to study entry. Except for curative skin basal cell carcinoma, carcinoma in situ or breast cancer >3 years.
2. Has received prior therapy with: anti-PD-1, anti-PD-L1, or anti-cytotoxic T-lymphocyte antigen 4 (CTLA-4) antibodies; Famitinib; patient is allergic to monoclonal antibody.
3. Known to have autoimmune disease.
4. Recived other anticancer therapy 4 weeks before randomization.
5. Known to be human immunodeficiency virus positive, active hepatitis B virus, or active hepatitis C virus.
6. Untreated and/or uncontrolled brain metastases.
7. With high risk of vaginal bleeding or gastrointestinal perforation.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) assessed by Blinded Independent Central Review in recurrent or metastatic cervical cancer patients(SHR-1210+Famitinib versus SHR-1210) | Up to approximately 2 years
  Defined as the number of subjects with a best overall response (BOR) of CR (Disappearance of all target lesions) or PR (At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) divided by the number of measurable subjects with target lesion at baseline according to RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Progression free survival (PFS) in recurrent or metastatic cervical cancer patients(SHR-1210+Famitinib versus SHR-1210) | Up to approximately 2 years
  PFS is defined as from the time of randomization until the date of first documented progression or date of death from any cause, whichever came first.
Overall survival (OS) in recurrent or metastatic cervical cancer patients(SHR-1210+Famitinib versus SHR-1210) | Up to approximately 2 years
  OS is the time interval from randomization to death due to any reason or lost of follow-up.
Objective Response Rate (ORR) assessed by investigator in recurrent or metastatic cervical cancer patients(SHR-1210+Famitinib versus SHR-1210) | Up to approximately 2 years
  Defined as the number of subjects with a best overall response (BOR) of CR (Disappearance of all target lesions) or PR (At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) divided by the number of measurable subjects with target lesion at baseline according to RECIST 1.1 criteria.
Disease control rate (DCR)，recurrent or metastatic cervical cancer patients(SHR-1210+Famitinib versus SHR-1210) according to RECIST 1.1 criteria | Up to approximately 2 years
  Defined as the number of subjects with a best overall response (BOR) of CR (Disappearance of all target lesions), PR (At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) or SD (Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.) divided by the number of measurable subjects with target lesion at baseline according to RECIST 1.1 criteria.
Duration of response (DoR), in recurrent or metastatic cervical cancer patients(SHR-1210+Famitinib versus SHR-1210) according to RECIST 1.1 criteria. | Up to approximately 2 years
  For participants who demonstrate CR or PR, DOR is defined as the time from first documented evidence of CR or PR until disease progression or death from any cause, whichever came first. The DOR per RECIST 1.1 as assessed by Investigator will be presented.
Time to response (TTR), in recurrent or metastatic cervical cancer patients(SHR-1210+Famitinib versus SHR-1210) according to RECIST 1.1 criteria. | Up to approximately 2 years
  Defined as the time from randomization to the first objective tumor response (At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters)) observed for patients who achieved a CR or PR.
Time to treatment failure (TTF)，in recurrent or metastatic cervical cancer patients(SHR-1210+Famitinib versus SHR-1210) according to RECIST 1.1 criteria. | Up to approximately 2 years
  Defined as the time from randomization to the end of treatment or death from any cause, whichever came first.
Adverse Events (AEs) | from the first drug administration to within 90 days for the last treatment dose
Tolerance | from the first drug administration to within 90 days for the last treatment dose
  To calculate the proportion of dose interruption, dose reduction or dose termination because of drug-related toxicity
Characteristic of Anti drug antibody | from the first drug administration to within 90 days for the last treatment dose
  Defined as ratio of ADAs of SHR-1210 during the treatment compared to baseline.
Peak Serum Concentration of SHR-1210 | from the first drug administration to within 90 days for the last treatment dose
  Defined as peak serum concentration of SHR-1210 during the treatment compared to baseline
Peak Plasma Concentration of famitinib | from the first drug administration to within 90 days for the last treatment dose
  Defined as peak plasma concentration of famitinib during the treatment compared to baseline
Area under the Serum Concentration versus Time Curve of SHR-1210 | from the first drug administration to within 90 days for the last treatment dose
  Defined as area under the serum concentration versus time curve of SHR-1210 during the treatment compared to baseline
Area under the Plasma Concentration versus Time Curve of famitinib | from the first drug administration to within 90 days for the last treatment dose
  Defined as area under the plasma concentration versus time curve of famitinib during the treatment compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xia L, Zhang K, Tang Y, Zhang G, Wang D, Lou H, Liu N, Zhang H, Chen H, Wang K, Wei S, Wang L, Gao K, Li G, Zhang H, Hu Y, Zhao W, Zhang Y, Zhu H, Lin A, Miao J, Yu G, Hua K, Tang L, Liu Z, Zhang B, Li H, Zheng M, Wang X, Li F, Yang X, Zhou H, Xia B, Zhou X, Wang Y, Wang Q, Wu X. Camrelizumab Plus Famitinib versus Camrelizumab Alone and Investigator's Choice of Chemotherapy in Recurrent or Metastatic Cervical Cancer: A Randomized, Phase II Study. J Clin Oncol. 2025 Aug 20;43(24):2720-2733. doi: 10.1200/JCO-24-02495. Epub 2025 Jun 25. PMID 40561369